CLINICAL TRIAL: NCT05604391
Title: The Effect of Two Different Graft Positioning Techniques on Creeping Attachment in Free Gingival Graft Operations
Brief Title: The Effect of Free Gingival Graft on Root Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berceste Guler (Other)
Responsible Party: Sponsor-Investigator, Berceste Guler, Associate Professor, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-02/09
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession; Lack of Keratinized Gingiva
Keywords: free gingival grafts; creeping attachment; root closure; gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Method clinical trial Free gingival graft application has been a routine and successful treatment option since the 1960s. Positioning methods are applied on or apical gingival recession. The aim of this study is to evaluate the effect of two different free gingival graft positioning techniques on the creeping attachment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free gingival grafts to be placed apical to the gingival recession. (Active Comparator): It is the application of free gingival graft to the apical part of the recession area of mandibular anterior teeth with gingival recession and keratinized gingival height deficiency.
  Interventions: Procedure: Free gingival graft placed apically
- Free gingival grafts to be placed coronal to the gingival recession. (Active Comparator): It is the application of free gingival graft to the coronal part of the recession area of mandibular anterior teeth with gingival recession and keratinized gingival height deficiency.
  Interventions: Procedure: Free gingival graft placed coronally

INTERVENTIONS:
Procedure: Free gingival graft placed apically — For free gingival graft operation, the recipient area will be prepared with a half-thickness flap. A graft with a thickness of approximately 1.5 mm and a width and height of the recipient bed will be obtained from the palatal region in accordance with the recipient bed, and it will be sutured by placing it in the apical region of the gingival recession according to the randomly selected positioning technique.
  Arms: Free gingival grafts to be placed apical to the gingival recession.
Procedure: Free gingival graft placed coronally — For free gingival graft operation, the recipient area will be prepared with a half-thickness flap. A graft with a thickness of approximately 1.5 mm and a width and height of the recipient bed will be obtained from the palatal region in accordance with the recipient bed, and it will be sutured by placing the coronal region of the gingival recession according to the randomly selected positioning technique.
  Arms: Free gingival grafts to be placed coronal to the gingival recession.

SUMMARY:
Free gingival graft is a mucogingival surgical technique applied to increase keratinized gingival width and reduce gingival recession. Free gingival graft is one of the most widely used approaches in root closure treatments and in increasing the height of the keratinized gingiva. Evaluation of the effect of the amount of creeping attachment on the root surface caused by the free gingival grafts placed coronally and apical to the mucogingival line on the gingival recession in the mandibular anterior region with keratinized gingival deficiency with gingival recession. Forty patients with gingival recession and insufficient keratinized gingival height will be randomly divided into 2 main groups as free gingival grafts to be placed coronal and apical to the gingival recession.

DETAILED DESCRIPTION:
Free gingival graft is a mucogingival surgical technique applied to increase keratinized gingival width and reduce gingival recession. Free gingival graft is one of the most widely used approaches in root closure treatments and in increasing the height of the keratinized gingiva. The "creeping attachment" phenomenon draws attention in the long-term success of root closure treatment in areas with gingival recession. "Creeping attachment" is defined as the coronal movement of the gingiva in the area where free gingival graft or connective tissue is applied in the postoperative period. The mean root closure rate with the creeping attachment is approximately 1 mm and can be detected 1 to 36 days after graft surgery. In the literature, clinical studies that measured a creeping attachment value between 0.12 and 3.5 mm in a 2-year period in free gingival grafts applied to the marginal gingival level have been reported.

Systemically healthy and non-smoking patients older than 18 years of age who applied to Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology and had gingival recession in mandibular anterior teeth and keratinized gingival deficiency will be included in the study. Systemic and dental anamnesis will be taken from the patient before the operation and clinical measurements will be recorded.

Patients will be divided into 2 main groups as free gingival grafts to be placed coronal and apical to the gingival recession. They will be written as Group I and Group II in sealed envelopes and apical and coronal positioning groups will be chosen randomly.

The operation date will be given after the patient is given oral hygiene training and 4 weeks after receiving Phase I routine periodontal treatment. The data to be obtained preoperatively and postoperatively are as follows:

Clinical measurements

1. Plaque index (Löe&Silness): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
2. Gingival index (Silness&Löe): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
3. Attachment loss: It is the value of the distance between a tooth and the free gingiva based on the enamel-cementum boundary measured using a periodontal sonde.
4. Bleeding index on probing (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual gingival parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
5. Pocket depth: It is the vertical distance measured between a standard periodontal probe and the base of the periodontal sulcus and the gingival margin.
6. Keratinized gingival height: It is the distance from the free gingival margin to the mucogingival junction line.
7. Keratinized gingival thickness: It is the distance measured between the gingival surface and hard tissue with a standard periodontal probe inserted perpendicular to the keratinized gingiva.
8. Gingival recession depth: It is obtained by measuring the distance between the gingival margin in the midbuccal region and the enamel-cementum boundary.
9. Gingival recession width: It is the mesio-distal width of the recession from the midpoint of the distance between the enamel cementum border and the gingival margin.
10. Gingival phenotype: Visibility of the periodontal tube in the sulcus
11. Vestibular sulcus depth: It is the distance measured from the gingival margin to the base of the sulcus.

Sample Selection: Taking the effect size of 0.08 for the significance value in the G Power analysis program as a reference to a previously presented study, 40 teeth were planned to be taken for α= 0.05 and 80% power.

Statistical Analysis method:

All analyzes will be done with SPSS software. Intra-group temporal evaluations in test and control groups will be evaluated using Pairedsample -T or Wilcoxon test according to normal distribution values. For intergroup comparisons, according to the normal distribution of data, Student-t test will be analyzed in parametric within-group evaluations and Mann Withney U test in nonparametrics. The normal distribution of the data will be evaluated with the Kolmogorov-Smirnov test. The significance value will be taken as 0.05. Relationships between variables will be evaluated with Logistic Regression Analysis or Multivariate Regression Analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-99 years old
2. The patient does not have any systemic disease
3. Presence of at least one tooth with gingival recession in the mandibular anterior region
4. Excessive dentin sensitivity and impaired esthetics associated with recession
5. Identification of the enamel-cementum boundary in the shrinkage region
6. The tooth is alive and there are no irregularities, grooves, caries and restorations in the area to be treated.
7. No periodontal surgical treatment in the relevant areas in the last 24 months
8. Presence of adequate keratinized and attached gingiva in the donor area

Exclusion Criteria:

1. Being outside the specified age range
2. Any contraindication for systematic periodontal surgery
3. Failure to define the enamel-cementum boundary in the withdrawal region
4. Presence of caries, restoration, root concavity in the area to be treated
5. Patients who smoke more than 10 cigarettes per day
6. Patients who use drugs that suppress the immune system or impair recovery
7. Patients using drugs that impair bleeding
8. Insufficient keratinized and attached gingiva in the donor area

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
1. Percent closure of the gingival recession | Postoperatively 1th month, Postoperatively 3th month, Postoperatively 6th month, Postoperatively 12th month
  It is calculated by dividing the pre- and post-surgical values of the exposed root surface.

SECONDARY OUTCOMES:
2. Keratinized mucosa width change | Postoperatively 1th month, Postoperatively 3th month, Postoperatively 6th month, Postoperatively 12th month
  It is the pre- and post-surgical variation of the distance from the free gingival margin to the mucogingival junction line.
3. Keratinized mucosa width thickness change | Postoperatively 1th month, Postoperatively 3th month, Postoperatively 6th month, Postoperatively 12th month
  It is the pre- and post-surgical variation of the distance measured between the gingival surface and hard tissue with a standard periodontal probe inserted perpendicular to the keratinized gingiva.
4. Vestibular sulcus depth change | Postoperatively 1th month, Postoperatively 3th month, Postoperatively 6th month, Postoperatively 12th month
  It is the pre- and post-surgical variation of the distance measured from the gingival margin to the base of the sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
ndividual participant data can be shared if the principal investigator is contacted
Supporting Information: CSR
Time Frame: Following acceptance of manuscript
Access Criteria: Individual participant data can be shared if the principal investigator is contacted

REFERENCES:
- [Background] Dorfman HS, Kennedy JE, Bird WC. Longitudinal evaluation of free autogenous gingival grafts. J Clin Periodontol. 1980 Aug;7(4):316-24. doi: 10.1111/j.1600-051x.1980.tb01974.x. PMID 6936409
- [Background] Agudio G, Nieri M, Rotundo R, Franceschi D, Cortellini P, Pini Prato GP. Periodontal conditions of sites treated with gingival-augmentation surgery compared to untreated contralateral homologous sites: a 10- to 27-year long-term study. J Periodontol. 2009 Sep;80(9):1399-405. doi: 10.1902/jop.2009.090122. PMID 19722789
- [Background] Bell LA, Valluzzo TA, Garnick JJ, Pennel BM. The presence of "creeping attachment" in human gingiva. J Periodontol. 1978 Oct;49(10):513-7. doi: 10.1902/jop.1978.49.10.513. PMID 282425
- [Background] Matter J, Cimasoni G. Creeping attachment after free gingival grafts. J Periodontol. 1976 Oct;47(10):574-9. doi: 10.1902/jop.1976.47.10.574. PMID 1067400
- [Background] Gul SS, Zardawi FM, Sha AM, Rauf AM. Assessment of Creeping Attachment after Free Gingival Graft in Treatment of Isolated Gingival Recession. J Int Acad Periodontol. 2019 Jul 1;21(3):125-131. PMID 31473705